CLINICAL TRIAL: NCT06459505
Title: Effects of Adapted Physical Activities in Children With Hemiplegic Cerebral Palsy
Brief Title: Adapted Physical Activities in Hemiplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0789
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: Cerebral Palsy, Hemiplegia , Adapted Physical Activities.
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia

STUDY DESIGN:
Intervention Model Description: Parallel Assignment It will be Randomized control trial in which non probabilty convenient sampling will be used. Two groups of 7-11 age will be formed in which participants will be randomly divided. Group A will Adapted Physical Activities and group B will only receive conventional Physical Therapy used for hemiplegic cerebral palsy.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine or standard Physical Therapy Group (Active Comparator): This group will receive routine or conventional physical therapy.
  Interventions: Other: Routine or standard Physical Therapy
- Adapted Physical Activity Group (Experimental): This group will receive Adapted Physical Activities.
  Interventions: Other: Adapted Physical Activity

INTERVENTIONS:
Other: Routine or standard Physical Therapy — Participants will undergo physical therapy to stop abnormal movement patterns and restore control over output in the developmental sequence. Therapists will provide cues to elicit basic posture and movement patterns, inhibiting aberrant patterns. The therapy aims to promote normal posture and movement patterns, incorporating the hemiplegic side for symmetry and functional use. Active usage and targeted strengthening activities will be emphasized, with motor performance practice included.
  Arms: Routine or standard Physical Therapy Group
Other: Adapted Physical Activity — For Upper extremities, Manual Ability Classification Scale (MACS) is a tool designed to support individuals with hemiplegic cerebral palsy by providing structured support through activities focusing on strength, flexibility, balance, and coordination. Participants at different MACS levels receive tailored treatments, including adaptive tools, task-specific training, assistive gadgets, and functional training. For lower extremities, the therapy will begin on stable support surfaces before progressing to more challenging surfaces such as inflatable cushions, foam pads, or balance discs, focusing on slow and controlled motions for improved body alignment and coordination.
  Arms: Adapted Physical Activity Group

SUMMARY:
The rehabilitation process is critical for people with disabilities, and it appears reasonable to predict that adaptive physical activity will become an important instrument for holistic development in a human rights perspective within an ecological framework. To highlight appropriate physical activity and emphasise its importance as a space for social expression while designing rehabilitation and social inclusion procedures, as well as determining what the lines are and how to approach them. Cerebral palsy (CP) refers to a group of mobility and posture abnormalities caused by non-progressive interference in the growing brain.

This randomised controlled trial will recruit patients using non-probability convenience sampling. Data will be gathered from the Pakistan Society of Rehabilitation Sciences (PSRD) and Behaviour and Special Education Services (BASES). Children diagnosed with hemiplegic cerebral palsy will be included. Patients will be placed into two groups: group 1 will receive an adapted physical activity program, while group 2 will receive conventional care/routine physical therapy. Both groups will receive 30-minute sessions per day, three days a week, for six weeks. The study will use pre- and post-test assessments of patients using the Manual Ability Classification Scale, Gross Motor Function Measure, Goal Attainment Scale, and Lower Extremity Functional Scale.The data will be analysed with SPSS version 25 software.

DETAILED DESCRIPTION:
GROUP A will receive pre-intervention evaluation that includes baseline measurements using the Manual Ability Classification Scale (MACS), Paediatric Evaluation of Disability Inventory (PEDI), Goal Attainment Scale (GAS), and Lower Extremity Functional Scale (LEFS) at 0 weeks.Participants will receive the modified physical activity program, the experimental group will take part. This program will involve adapted exercises, physical therapy, or modified sports, all aimed at meeting the unique requirements and difficulties faced by people with hemiplegic cerebral palsy and will help them improve their dynamic balance, equilibrium, strength and flexibility. Daily video recordings will be used to collect feedback. Mothers will participate in therapy sessions. Utilizing appropriate assessment instruments and outcome measures, the experimental group's advancement and results will be continuously observed and evaluated. For upper extremity participants will be categorized according to their the MACS level. The levels range from I (able to handle objects easily) to V (limited ability to handle objects). Interventions should be individualized based on the specific needs identified through the MACS assessment. The levels go from I, which is an easy level of object handling, to V, which is a limited degree of object handling. Individualized interventions should be developed in accordance with the unique needs that the MACS evaluation has revealed. Treatment session of 30 minutes per day for three days a week, for six weeks for each participant. After that post-test assessment will be conducted through MACS, PEDI, GAS and LEFS.

Group B will have regular therapy or conventional care that is normally given to people with hemiplegic cerebral palsy. The same evaluation instruments and outcome measures that are used for the experimental group will also be used for the control group's monitoring and assessment. Each participant will receive 30 minutes of treatment three days per week for 6 weeks, spread out over four days of the week. Following that, post-test evaluations using MACS, PEDI, GAS, and LEFS will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemiplegic cerebral palsy who have been diagnosed fall within the age range of 7 to 11 years.
* GMFCS will be hired at the I-II level.
* Individuals with steady health conditions

Exclusion Criteria:

* Diseases or traumas that would make physical therapy inappropriate or dangerous.
* Have previously engaged in a comparable program for adaptive physical activity
* Leave out kids who have recently had Botox injections
* Inability to commit to the study protocol or attend scheduled therapy sessions

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Manual Classification Scale of Ability (MACS) | 6 weeks
  This tool was created to categorise people with cerebral palsy according to their manual abilities. Based on an individual's self-initiated ability to handle objects, it offers a five-level rating system that emphasises hand use throughout daily activities. Reliability between tests; r = (ICC = 0.984). Mini-MACS and the Gross Motor Function Classification System were found to be correlated (r = 0.626, 0.596, and 0.598)
Pediatric Evaluation of Disability Inventory (PEDI) | 6 weeks
  Use of the Pediatric Evaluation of Disability Inventory (PEDI): This assessment tool assesses children with impairments' performance and functional abilities. Researchers, therapists, and healthcare professionals frequently utilize the PEDI to evaluate a child's abilities in a variety of daily life domains. ICC = 0.845-0.938, Cronbach's alpha = 0.889-0.964
Goal Attainment Scale (GAS) | 6 weeks
  An outcome measure intended to evaluate how well people accomplish their objectives over the course of a given intervention or treatment period. It is frequently employed in several industries, such as healthcare, education, and rehabilitation. GAS is a versatile instrument in evaluating progress towards customised targets since it enables the individualization of goal setting and outcome evaluation. Reliability between and within testers (ICC=0.98)
Lower Extremity Functional Scale (LEFS): | 6 weeks
  Frequently use to evaluate the functional status of patients with musculoskeletal disorders of the lower extremities. It is frequently used to gauge a person's capacity for carrying out different tasks linked to lower limb function in orthopaedic and physical therapy settings. The LEFS often asks about a person's capacity for carrying out routine tasks including running, jumping, walking, and stair climbing. The overall functional status of the lower extremities is assessed using the ratings that respondents provide on a scale for each activity. Intraclass correlation values (ICC=0.85-0.99) and Pearson correlation=(>0.7)

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Mangrio, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab, Pakistan, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sit C, Aubert S, Carty C, Silva DAS, Lopez-Gil JF, Asunta P, Palad Y, Guisihan R, Lee J, Arbour Nicitopoulos KP, Vanderloo LM, Stanish H, Haegele J, Urbanski PK, Pozeriene J, Hutzler Y, Ng K. Promoting Physical Activity Among Children and Adolescents With Disabilities: The Translation of Policy to Practice Internationally. J Phys Act Health. 2022 Oct 22;19(11):758-768. doi: 10.1123/jpah.2022-0351. Print 2022 Nov 1. PMID 36280232